CLINICAL TRIAL: NCT06500247
Title: A Prospective Exploratory Phase II Study on the Treatment of Advanced Metastatic Castration-resistant Prostate Cancer With Darxicilib in Combination With Abiraterone Acetate (II)
Brief Title: Darxicilib Combined With Abiraterone Acetate Tablets (II) for the Treatment of Advanced Metastatic Castration-resistant Prostate Cancer.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: bks04
Record Dates: First submitted 2024-06-27; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-06

CONDITIONS: The Efficacy of Abiraterone Acetate Combined With Dalpicilib in the Treatment of Patients With Metastatic Castration-resistant Prostate Cancer
Keywords: Prostate Cancer; CDK4/6 inhibitor; Abiraterone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Androgen Antagonists; Prednisone

STUDY DESIGN:
Intervention Model Description: Experimental group:Dalpicilib+Abiraterone Acetate (II) +ADT+Prednisone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Androgen Deprivation Therapy+Darxicilib+Abiraterone Acetate（II）+Prednisone
  Interventions: Drug: Dalpicilib; Drug: Abiraterone Acetate (II); Drug: Androgen Deprivation Therapy; Drug: Prednisone

INTERVENTIONS:
Drug: Dalpicilib — This study recruited a total of 43 subjects diagnosed with Metastatic Castration-Resistant Prostate Cancer at multiple centers from July 2024. Enrolled patients received treatment with dalpicilib until disease progression or intolerable toxicity, with a maximum treatment duration of up to 2 years. Follow-up visits were conducted monthly after patient enrollment. The last follow-up was completed in March 2027.
Drug: Abiraterone Acetate (II) — This study recruited a total of 43 subjects diagnosed with Metastatic Castration-Resistant Prostate Cancer at multiple centers from July 2024. Enrolled patients received treatment with Abiraterone Acetate (II) until disease progression or intolerable toxicity, with a maximum treatment duration of up to 2 years. Follow-up visits were conducted monthly after patient enrollment. The last follow-up was completed in March 2027.
Drug: Androgen Deprivation Therapy — This study recruited a total of 43 subjects diagnosed with mCRPC at multiple centers from July 2024. Enrolled patients received treatment with Androgen Deprivation Therapy until disease progression or intolerable toxicity, with a maximum treatment duration of up to 2 years. Follow-up visits were conducted monthly after patient enrollment. The last follow-up was completed in March 2027.
Drug: Prednisone — This study recruited a total of 43 subjects diagnosed with mCRPC at multiple centers from July 2024. Enrolled patients received treatment with Prednisone until disease progression or intolerable toxicity, with a maximum treatment duration of up to 2 years. Follow-up visits were conducted monthly after patient enrollment. The last follow-up was completed in March 2027.

SUMMARY:
This study is a single-arm, multicenter, phase II exploratory trial. The purpose is to explore the efficacy and safety of Darxicilib in combination with Abiraterone Acetate for the treatment of subjects with metastatic castration-resistant prostate cancer.The main questions it aims to answer are:

·PSA50 response rate at the end of week 12

Participants will:

* Darxicilib: 125mg per tablet, oral administration, once daily for 21 consecutive days followed by a 7-day break.
* Abiraterone Acetate tablets (II): 300mg per dose, oral administration, once daily for a 28-day cycle.
* Prednisone: 5mg per tablet, oral administration, twice daily.

DETAILED DESCRIPTION:
1. This research constitutes a phase II, single-arm, multicenter exploratory study aimed at assessing the therapeutic efficacy and safety profile of the combination therapy involving Darxicilib and Abiraterone Acetate (II) in patients diagnosed with metastatic castration-resistant prostate cancer (mCRPC). The enrollment target is set at 43 participants who meet the eligibility criteria for the efficacy assessment phase of the trial.
2. (1)Main Research Objective To evaluate the efficacy of the treatment modality of Darxicilib in combination with Abiraterone Acetate (II) in patients with mCRPC (metastatic castration-resistant prostate cancer).

(2)Secondary Research Objectives

1. To assess the efficacy of the combination therapy in target mCRPC subjects through the time to PSA progression, PSA response rate at 12 weeks (PSA50, PSA90, and PSA ≤ 0.2 ng/ml), disease-free survival (PFS) rates at 6 and 12 months, overall survival (OS), and duration of response (DOR);
2. To evaluate the safety of the combination therapy for target mCRPC by assessing the incidence of adverse events, time to pain progression, and time to symptom progression.

(3)Exploratory Research Objective Quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old, male;
* ECOG performance status score of 0 to 1;
* Life expectancy of at least 3 months;
* Histologically or cytologically confirmed adenocarcinoma of the prostate, without a diagnosis of neuroendocrine or small cell carcinoma;
* Testosterone at castrate levels at screening (≤50 ng/dL or 1.73 nmol/L);
* Failure of previous treatment with new androgen receptor antagonists at the mHSPC stage (such as enzalutamide, apalutamide, ODM-201, SHR3680, HC-1119, and pucrol);
* Capable of complying with the study protocol as judged by the investigator;

Exclusion Criteria:

* Previously received abiraterone acetate treatment for prostate cancer;
* Previously received any cytotoxic chemotherapy for mCRPC stage;
* Previously received treatment with any other cyclin-dependent kinase 4 and 6 (CDK4 & 6) inhibitors;
* Previously received treatment with new androgen receptor antagonists at the mCRPC stage (such as enzalutamide, apalutamide, ODM-201, SHR3680, HC-1119, and pucrol);
* The washout period from the end of any previous anti-tumor treatment (including radiotherapy, surgery, molecular targeted therapy, immunotherapy, and first-generation androgen receptor antagonists) to the first administration of this study is less than 4 weeks (except for bicalutamide with a washout period less than 6 weeks);

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2024-07-31 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
12 Week PSA 50 | 12 weeks
  Response rate of PSA 50 at the end of 12 weeks.

SECONDARY OUTCOMES:
Radiographic Progression-Free Survival | 3 years
  The time from randomization until the occurrence of radiographic progression or death from any cause.
Adverse event | 3 years
  During the trial, adverse events are assessed based on laboratory and clinical examinations.
overall survival | 3 years
  The time from the start of the study or the initiation of treatment for the patient, to the time of death from any cause.
PSA 50 | 3 years
  PSA 50 is defined as the percentage of patients experiencing a reduction in prostate-specific antigen (PSA) levels by at least 50% from their baseline values after treatment.
PSA 90 | 3 years
  PSA 90 is defined as the percentage of patients experiencing a reduction in prostate-specific antigen (PSA) levels by at least 90% from their baseline values after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No